CLINICAL TRIAL: NCT03033160
Title: A Randomized Controlled Trial of Vaginal Estrogen to Treat Asymptomatic Microscopic Hematuria
Brief Title: Vaginal Estrogen for Asymptomatic Microscopic Hematuria
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Boston Urogynecology Associates (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Mount Auburn Hospital (Other)
Responsible Party: Principal Investigator, Lekha S. Hota, Clinical Instructor Division of Urogynecology and Female Pelvic Medicine and Reconstructive Surgery, Boston Urogynecology Associates
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 052-2015
Record Dates: First submitted 2016-10-19; First posted 2017-01-26 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Asymptomatic Microscopic Hematuria
Keywords: Estrogen; Hematuria
MeSH Terms: conditions — Hematuria | interventions — Estradiol

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Estradiol Ring (Experimental): Estradiol Ring per vagina every 3 months
  Interventions: Drug: Estradiol Ring
- Observation (No Intervention): Observation

INTERVENTIONS:
Drug: Estradiol Ring
  Other Names: Estring
  Arms: Estradiol Ring

SUMMARY:
The specific aim of this protocol is to determine whether vaginal estrogen is an effective treatment for asymptomatic microscopic hematuria in postmenopausal women. The investigators hypothesize that women who use vaginal estrogen for three months will be more likely to have resolution of their asymptomatic microscopic hematuria compared with women who do not use vaginal estrogen.

DETAILED DESCRIPTION:
This is a multi-center, randomized controlled trial to evaluate whether vaginal estrogen is an effective treatment for asymptomatic microscopic hematuria. Postmenopausal women with asymptomatic microscopic hematuria will be recruited from the two urogynecology clinics that serve as the clinic sites for the Mount Auburn Hospital/Beth Israel Deaconess Medical Center Female Pelvic Medicine and Reconstructive Surgery fellowship.

Participants are eligible if they are postmenopausal, defined by amenorrhea for at least one year or a bilateral oophorectomy at least one year prior, and have three or more red blood cells per high powered field visible in a properly collected urine specimen without evidence of infection. In addition, participants must have a negative cystoscopy and computed tomography urogram (or magnetic resonance urography if history of renal insufficiency or contrast allergy) within the past three years. Exclusion criteria include any of the following: current or past thromboembolic disorder or cerebrovascular accident, intolerance to previous estrogen replacement therapy or hormone replacement therapy, estrogen dependent neoplasm within the past five years (unless supporting documentation from patient's oncologist is obtained), estrogen replacement therapy or hormone replacement therapy within the past three months or selective estrogen receptor modulators within eight weeks of enrollment, urinary tract infection, urinary calculi, urinary tract malignancy, vaginal bleeding of unknown origin, urethral caruncle, history of recurrent urinary tract infections in the last one year, and stage two or greater pelvic organ prolapse.

Participants will be randomized to either an estradiol-releasing vaginal ring (Estring; Pfizer, New York, NY) or expectant management in a ratio of 1:1 using computer-generated block randomization stratified by enrollment site.

Estring is a silicone vaginal ring, 5.5 cm in diameter, containing 2 mg of 17-estradiol, which is released at a rate of 7.5 g daily. The Estring was chosen as the vehicle for vaginal estrogen secondary to its ease of administration, higher patient preference, acceptability, and compliance.

After eligibility is confirmed and written, informed consent is obtained, participants will be randomized to one of the two study arms. Participants randomized to the use of vaginal estrogen will have the vaginal ring placed by one of the investigators. Participants in both study arms will complete the short form of the Urogenital Distress Inventory (UDI-6) and the Incontinence Impact Questionnaire (IIQ-7).

Participants in the vaginal estrogen arm will be called at two, four and eight weeks to ensure that the Estring is still in place and follow-up appointments will be scheduled as needed if there is any question as to whether the ring is still in place.

At the 12-week visit all participants will provide a urine sample for urinalysis to assess whether the microscopic hematuria is present. All participants also will be asked to complete the UDI-6 and IIQ-7 and vaginal mucosal atrophy will be assessed as described above. Women in the vaginal estrogen arm will have the Estring removed and a new Estring will be placed by one of the investigators; participants also will be asked if the ring was removed or fell out during the past 12 weeks. All participants will be asked whether any of the following, (which could be a side effect from vaginal estrogen use) occurred in the previous 12 weeks: dyspareunia for subject or partner, vaginal bleeding, non-physiologic discharge, vaginal ulceration and vaginal irritation.

participants will be followed for 24 weeks to determine if more than 12 weeks are needed for resolution.

At the 24-week visit, all participants will provide a urine sample for urinalysis to assess whether the microscopic hematuria is present. All participants also will be asked to complete the UDI-6 and IIQ-7 and vaginal mucosal atrophy will be assessed as described above. We will ask all participants whether any of the following, which could be a side effect from vaginal estrogen use, occurred in the previous 12 weeks: dyspareunia for subject or their partner, vaginal bleeding, non-physiologic discharge, vaginal ulceration and vaginal irritation. One of the investigators will remove the Estring from all women in the vaginal estrogen arm.

At the 24 week visit investigators will offer women in the expectant management arm with persistent microscopic hematuria the opportunity to try the Estring.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, defined by amenorrhea for at least one year or a bilateral oophorectomy at least one year prior, and have three or more red blood cells per high powered field visible in a properly collected urine specimen without evidence of infection. In addition, women must have a negative cystoscopy and computed tomography urogram (or magnetic resonance urography if history of renal insufficiency or contrast allergy) within the past three years.

Exclusion Criteria:

* Current or past thromboembolic disorder or cerebrovascular accident
* Intolerance to previous estrogen replacement therapy or hormone replacement therapy
* Estrogen dependent neoplasm within the past five years (unless supporting documentation from patient's oncologist is obtained)
* Estrogen replacement therapy or hormone replacement therapy within the past three months or selective estrogen receptor modulators within eight weeks of enrollment
* Urinary tract infection
* Urinary calculi
* Urinary tract malignancy
* Vaginal bleeding of unknown origin
* Urethral caruncle
* History of recurrent urinary tract infections in the last one year
* Stage two or greater pelvic organ prolapse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-10 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of microscopic hematuria (RBC's) at 12 weeks compared to baseline measurement | 12 weeks
  Investigators will compare red blood cell count results obtained during the initial urinalysis to the 12 week urinalysis to measure any change in red blood cell count (if any).

SECONDARY OUTCOMES:
Comparison of Microscopic Hematuria (RBC's) at 24 weeks compared to baseline. | 24 weeks
  Investigators will cimpare red blood cell count results obtained during the initial Urinalysis to the 24 week urinalysis to measure any change in red blood cell count (if any).
To Assess Quality of Life | 12 weeks
  Measurement of quality of life change from baseline, utilizing subject self administered questionnaires, Urogenital Distress Inventory Short Form (UDI-6) and the Incontinence Impact Questionnaire-short Form (IIQ-7)

CONTACTS AND LOCATIONS:
Overall Officials: Lekha Hota, MD, Principal Investigator — Practitioner
Locations (1):
- Mount Auburn Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No